CLINICAL TRIAL: NCT02344862
Title: Exploratory Study of FYU-981 for Hyperuricemia With or Without Gout (Phase II (IIa) Study)
Brief Title: Study of FYU-981 in Hyperuricemia With or Without Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FYU-981-003
Record Dates: First submitted 2015-01-18; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — dotinurad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- FYU-981 High dose (Active Comparator)
  Interventions: Drug: FYU-981 High dose, (Oral daily dosing for 8 weeks)
- FYU-981 Middle dose (Active Comparator)
  Interventions: Drug: FYU-981 Middle dose, (Oral daily dosing for 8 weeks)
- FYU-981 Low dose (Active Comparator)
  Interventions: Drug: FYU-981 Low dose, (Oral daily dosing for 8 weeks)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo, (Oral daily dosing for 8 weeks)

INTERVENTIONS:
Drug: FYU-981 High dose, (Oral daily dosing for 8 weeks) — Subjects randomized to the FYU-981 High dose arm receive active drug, FYU-981 High dose.
  Arms: FYU-981 High dose
Drug: FYU-981 Middle dose, (Oral daily dosing for 8 weeks) — Subjects randomized to the FYU-981 Middle dose arm receive active drug, FYU-981 Middle dose.
  Arms: FYU-981 Middle dose
Drug: FYU-981 Low dose, (Oral daily dosing for 8 weeks) — Subjects randomized to the FYU-981 Low dose arm receive active drug, FYU-981 Low dose.
  Arms: FYU-981 Low dose
Drug: Placebo, (Oral daily dosing for 8 weeks) — Subjects randomized to the placebo arm receive placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is exploratory investigation of safety and efficacy (dose response and optimal dose according to the percent reduction from baseline in serum urate level at the final visit) of FYU-981 administered orally to hyperuricemic patients with and without gout for 8 weeks (dose-escalating initial period: 4 weeks followed by maintenance period: 4 weeks) by the method of randomized (dynamic allocation), placebo-controlled, double-blind, parallel group comparison.

ELIGIBILITY:
Inclusion Criteria:

* Hyperuricemic or gout patients
* Serum urate level:

>= 7.0mg/dL in patients with history of gout, or >= 8.0mg/dL in patients with hypertension, diabetes or metabolic syndrome, or >= 9.0mg/dL

Exclusion Criteria:

* Gouty arthritis within two weeks before start of study treatment
* Secondary hyperuricemia
* HbA1c: >= 8.4%
* Uric acid-overproduction type in the classification of hyperuricemia
* History of, clinically significant cardiac, hematologic and hepatic disease
* Kidney calculi or clinically significant urinary calculi
* eGFR: < 60mL/min/1.73m^2
* Systolic blood pressure: >= 180 mmHg
* Diastolic blood pressure: >= 110 mmHg

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percent reduction from baseline in serum urate level at the final visit | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Tokyo, Japan

REFERENCES:
- [Derived] Hosoya T, Sano T, Sasaki T, Fushimi M, Ohashi T. Clinical efficacy and safety of dotinurad, a novel selective urate reabsorption inhibitor, in Japanese hyperuricemic patients with or without gout: an exploratory, randomized, multicenter, double-blind, placebo-controlled, parallel-group early phase 2 study. Clin Exp Nephrol. 2020 Mar;24(Suppl 1):44-52. doi: 10.1007/s10157-019-01802-w. Epub 2019 Nov 21. PMID 31754882